CLINICAL TRIAL: NCT04550507
Title: Mind-Body Interventions to Mitigate Effects of Media Use on Sleep (Sleepazoid Study)
Brief Title: Mind-Body Interventions to Mitigate Effects of Media Use on Sleep in Early Adolescents
Acronym: Sleepazoid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Michelle Garrison, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001443; R61AT009859 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-09-16 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Mindful Sensory Awareness (Experimental): Group A: Mindful Sensory Awareness receives the mindful sensory awareness intervention during the first 8-week period, and receives no active intervention delivery during the second 8-week period.
  Interventions: Behavioral: Mindful sensory awareness intervention
- Group B: Mindful Sensory and Body Awareness (Other): Group B: Mindful Sensory and Body Awareness receives no active intervention delivery during the first 8-week period, and during the second 8-week period receives an intervention combining the mindful sensory awareness content received by Group A with the mindful body awareness check-in approach.
  Interventions: Behavioral: Mindful sensory awareness + mindful body awareness check-ins intervention

INTERVENTIONS:
Behavioral: Mindful sensory awareness intervention — The mindfulness sensory awareness exercise will be a brief (3-5 minutes), guided meditation focusing on sensory and interoceptive awareness developed by Co-I Price, modified slightly to meet the needs of this age group and targeted for attention to indicators of fatigue or a sense of overstimulation. Youth will be asked to use the exercise after ending media use but before trying to sleep. The meditation component will be delivered via an audio-guided MP3, along with illustrated instructions in both handout and video, and a guided workbook that coaches youth over the 8-week intervention period to practice their skills, reflect on their experiences, and maintain adherence.
  Arms: Group A: Mindful Sensory Awareness
Behavioral: Mindful sensory awareness + mindful body awareness check-ins intervention — During the intervention period for Group B: Mindful Sensory & Body Awareness(the second 8 weeks), they will receive the same mindful sensory awareness intervention, and also learn the mindful body awareness check-ins to guide media use choices strategy (referred to here as the check-ins component). We will coach youth to pause briefly every 30 minutes during media use to discern if they detect physical, cognitive, or emotional signs of escalated state arousal, and to make an intentional and real-time choice about possible changes in media use content or duration to help decrease state arousal levels before bed.
  Arms: Group B: Mindful Sensory and Body Awareness

SUMMARY:
Eliminating media use is neither feasible at a public health level nor perhaps even desirable given the role it plays in the lives of youth and adults, but mind-body interventions have the potential to mitigate state arousal effects and thus reduce negative impacts on sleep. Given emerging literature on links between intensive media use, sensory and interoceptive awareness, and self-regulation, this study will examine two related mind-body approaches -- a mindfulness sensory awareness exercises and mindful body awareness check-ins -- in a randomized clinical trial of early adolescents with evening media use and sleep problems.

ELIGIBILITY:
Inclusion Criteria:

* Child age at enrollment is 11y0m to 14y11m
* Child is in the 6th-8th grade, or during summer recruitment, will be so in the coming autumn.
* Total score of 52 or higher on the Sleep Disturbances Scale for Children (SDSC), a parent-report survey questionnaire regarding child sleep health
* Parent reports child has >= 1 hour of media use during the 3 hours before bed at least 4 nights per week.
* Parent and child both are comfortable reading and hearing instructions in English and in answering surveys written in English.
* Families must also have at least two internet-connected portable screen devices available - one which much be an iOS or Android tablet or smartphone device and which will be used to download the games used in the media-induced arousal task and then used to play those games with the device in airplane mode, and a second which will be used to connect to the study staff via video conference, and which can be a laptop computer, tablet, or smartphone.

Exclusion Criteria:

* Untreated diagnosis (by parent report) or positive screen for sleep-disordered breathing on the SDSC parent report survey questionnaire
* Current use of medications known to affect sleep (systemic corticosteroids, stimulants, melatonin) by parent report
* Sleeps at a second residence from enrolling parent more than two nights a week according to parent report
* Has a current serious chronic medical condition known to affect sleep and/or arousal patterns (such as cancer or diabetes) by parent report.
* Currently engages in meditation or body scan to fall asleep, according to parent report

We exclude potential participants who meet one of the following criteria because of concerns that their heart rate variability response may be too atypical to be valuable in this protocol (ASD or developmental delay, eating disorder, PTSD, illicit drug use) and/or because of concerns that the associated behavioral challenges and/or instability would impair ability to adhere to the entire 4-6 month protocol.

* Diagnosis of Autism Spectrum Disorder or developmental delay by parent self-report
* Current diagnosis of eating disorder by parent self-report
* Current diagnosis of PTSD by parent self-report
* Illicit drug use within the last three months by parent self-report
* Is currently suicidal, based on the ASQ (Ask Suicide Screening Questions)
* Hospitalization for depression or anxiety in the last year by parent self-report; or severe current depression symptoms as indicated by a t-score > 80 on the RCADS-25. We will also exclude those with last year hospitalization, regardless of symptom score, because this is often an indicator of instability and undertreatment, and ability to adhere to the entire 4-6 month protocol would likely be impaired.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
state arousal measured by heart rate variability (HRV), 30 minutes prior to usual bedtime | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  HRV will be captured by wireless telemetry (Empatica E4 and Actiheart), and primary metrics will be the pNN50 (the proportion of successive pairs of beat-to-beat intervals differing by more than 50ms in length) and the RMSSD (the root mean square of successive differences across successive pairs of beat-to-beat intervals).
  HRV will be compared between intervention and control and operationalized as the median of the statistic over 5-minute time periods on each of the two measurement nights beginning at 30 minutes prior to usual bedtime.
state arousal measured by heart rate variability (HRV), beginning at usual bedtime | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  HRV will be captured by wireless telemetry (Empatica E4 and Actiheart), and primary metrics will be the pNN50 (the proportion of successive pairs of beat-to-beat intervals differing by more than 50ms in length) and the RMSSD (the root mean square of successive differences across successive pairs of beat-to-beat intervals).
  HRV will be compared between intervention and control and operationalized as the median of the statistic over 5-minute time periods on each of the two measurement nights beginning at usual bedtime.
state arousal measured by heart rate variability (HRV), when youth started trying to fall asleep | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  HRV will be captured by wireless telemetry (Empatica E4 and Actiheart), and primary metrics will be the pNN50 (the proportion of successive pairs of beat-to-beat intervals differing by more than 50ms in length) and the RMSSD (the root mean square of successive differences across successive pairs of beat-to-beat intervals).
  HRV will be compared between intervention and control and operationalized as the median of the statistic over 5-minute time periods on each of the two measurement nights beginning when the youth reported on the diary starting to try to fall asleep.
state arousal measured by heart rate variability (HRV), during game play exposure | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  HRV will be captured by wireless telemetry (Empatica E4 and Actiheart), and primary metrics will be the pNN50 (the proportion of successive pairs of beat-to-beat intervals differing by more than 50ms in length) and the RMSSD (the root mean square of successive differences across successive pairs of beat-to-beat intervals).
  HRV will be compared between intervention and control and operationalized as the median of the statistic over 5-minute time periods during the remote assessment visit during the last 5 minutes of the game play exposure.
state arousal measured by heart rate variability (HRV), during recovery period | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  HRV will be captured by wireless telemetry (Empatica E4 and Actiheart), and primary metrics will be the pNN50 (the proportion of successive pairs of beat-to-beat intervals differing by more than 50ms in length) and the RMSSD (the root mean square of successive differences across successive pairs of beat-to-beat intervals).
  HRV will be compared between intervention and control and operationalized as the median of the statistic over 5-minute time periods during the remote assessment visit during the last 5 minutes of the recovery period post-exposure.

SECONDARY OUTCOMES:
state arousal measured by electrodermal activity (EDA) | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  The Empatica E4 wrist-worn wireless telemetry device also measures electrodermal activity (EDA) in µSiemens, sampled at 4Hz. EDA will be compared between intervention and control and operationalized as the median of the statistic over 5-minute time periods per measurement night at each of the following time periods, both in the home measurement weeks: a) beginning at 30 minutes prior to usual bedtime, b) beginning at usual bedtime, and c) beginning when the youth reported starting to try to fall asleep, with (b) and (c) being further apart on nights with greater behavioral bedtime delay, and in the remote assessments: d) in the last 5 minutes of the game play exposure, and e) in the last 5 minutes of the recovery period post-exposure.
PreSleep Arousal Scale, modified for Children (PSAS-C), remote assessment visits | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  The PSAS-C (PreSleep Arousal Scale, modified for Children) is a 16-item scale that has been successfully used to assess perceived cognitive and somatic arousal at bedtime in children ages 8-14; and the adult version (PSAS) has been shown to be a significant mediator of the relationship between evening media use and sleep in adolescents and young adults, and been used to test state arousal mechanisms of mindfulness interventions on sleep. Youth will complete this at the end of the post-exposure recovery period during each remote assessment visit. Possible scores range from 16-80, with higher scores indicating worse pre-sleep arousal levels.
PreSleep Arousal Scale, modified for Children (PSAS-C), home measurement weeks | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  The PSAS-C (PreSleep Arousal Scale, modified for Children) is a 16-item scale that has been successfully used to assess perceived cognitive and somatic arousal at bedtime in children ages 8-14; and the adult version (PSAS) has been shown to be a significant mediator of the relationship between evening media use and sleep in adolescents and young adults, and been used to test state arousal mechanisms of mindfulness interventions on sleep. Youth will complete this each night during all home measurement weeks as part of the sleep diary, and the mean result across the week will be used. Possible scores range from 16-80, with higher scores indicating worse pre-sleep arousal levels.
mean sleep onset latency (SOL) | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  time from diary-reported "going to bed" time to diary-reported time of sleep onset, averaged across one week
mean sleep duration | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  diary-reported time of sleep onset to diary-reported time of sleep offset, averaged across one week
Adolescent Sleep Wake Scale (ASWS) total sleep scale score | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  The ASWS (Adolescent Sleep Wake Scale) is a symptom scale of behavioral sleep problems common across pre-adolescence and adolescence, chosen because it does not focus on school days (and so appropriate year-round) and is written at Flesch-Kincaid Grade 4.5. Possible scores range from 5-30, with higher scores indicating better sleep.
time to reach baseline arousal (HRV and EDA) | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  We will also evaluate the time to reach baseline state arousal levels (via HRV and EDA) after ceasing evening media use will be decreased in the intervention compared to the control group, in both remote assessment visit and home measurement week settings.

OTHER OUTCOMES:
Adolescent Sleep Hygiene Scale (ASHS) total sleep hygiene score | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  The ASHS (Adolescent Sleep Hygiene Scale) is a scale measuring environmental and behavioral factors contributing to sleep problems common across pre-adolescence and adolescence, chosen because it does not focus on school days (and so appropriate year-round) and is written at Flesch-Kincaid Grade 4.5. It is collected via youth self-report surveys. Possible scores range from 8-48, with higher scores indicating better sleep hygiene.
Cleveland Adolescent Sleepiness Questionnaire (CASQ) | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  Survey instrument to measure excessive daytime sleepiness in adolescent, collected via youth self-report surveys. Possible scores range from 0-80, with higher scores indicating worse daytime sleepiness.
MAIA-2 | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  This is a tool for evaluating interoceptive awareness, with subscales for noticing body sensations, attention regulation to body sensations, awareness of emotion signals in body sensations, etc. It is collected via youth self-report surveys. Possible scores range from 0-40, with higher scores indicating greater levels of positive awareness.
Revised Child Anxiety and Depression Scale, short form (RCADS-25) | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  This is a survey tool for assessing parent and youth report of anxiety and depression symptoms in the youth, collected via youth self-report surveys. Possible scores range from 0-75, with higher scores indicating more severe levels of anxiety and depression symptoms.
average screentime blackout | At baseline, and then at 8-12 weeks (directly after subjects complete intervention period A), and then at 16-20 weeks (directly after subjects complete intervention period B).
  This will be measured as the average time across a diary week at which a youth discontinued media use for the night. If the youth fell asleep while using media use, the time of sleep onset is used.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Garrison, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States